CLINICAL TRIAL: NCT02354482
Title: Achieving Patient-Centered Care and Optimized Health In Care Transitions by Evaluating the Value of Evidence
Acronym: ACHIEVE
Status: Completed | Type: Observational
Sponsor: Mark Williams (Other)
Collaborators: University of Pennsylvania (Other); Boston Medical Center (Other); Westat (Other); Kaiser Permanente (Other); Telligen, Inc. (Industry); University of Illinois at Chicago (Other); Hospital Research & Education Trust, American Hospital Association (Unknown); Joint Commission Resources (Unknown); America's Essential Hospitals (Other); Louisiana State University Health Sciences Center Shreveport (Other); United Hospital Fund (Other); Caregiver Action Network (Unknown); National Association of Area Agencies on Aging (Unknown)
Responsible Party: Sponsor-Investigator, Mark Williams, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 3048112229
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Care Transitions
MeSH Terms: interventions — Restraint, Physical; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diverse, high-risk patient populations
  Interventions: Behavioral: Patient Communication and Care Management; Behavioral: Home-Based Trust, Plain Language, and Coordination; Behavioral: Hospital-Based Trust, Plain Language, and Coordination; Behavioral: Patient/Caregiver Assessment and Provider Information Exchange; Behavioral: Assessment and Teach Back; Other: Standard of Care (Reference)

INTERVENTIONS:
Behavioral: Patient Communication and Care Management — Received the following Transitional Care strategies:
  1. Helpful Health Care Contact OR Symptom Management
  2. Post-discharge Care Consultation
  3. Patient Goal/Preference Assessment
  4. Plain Language Communication in Hospital
  5. Plain Language Communication at Home
  6. Transition Summary for Patients and Family Caregivers
Behavioral: Home-Based Trust, Plain Language, and Coordination — Received the following Transitional Care Strategies:
  1. Transition Team
  2. Home visits
  3. Plain Language Communication at Home
  4. Promote Trust at Home
  5. Referral to Community Services
  6. Follow-up Appointment
Behavioral: Hospital-Based Trust, Plain Language, and Coordination — Received the following Transitional Care Strategies:
  1. Post-discharge care consultation
  2. Identify High-Risk Patients and Intervene
  3. Medication Reconciliation
  4. Plain Language Communication in Hospital
  5. Promote Trust in the Hospital
  6. Transition Summary for Patients and Family Caregivers
Behavioral: Patient/Caregiver Assessment and Provider Information Exchange — Received the following Transitional Care Strategies:
  1. Patient Goal/Preference Assessment
  2. Identify High-Risk Patients and Intervene
  3. Timely Exchange of Critical Patient Information among Providers
  4. Patient/Family Caregiver Transitional Care Needs Assessment
Behavioral: Assessment and Teach Back — Received the following Transitional Care Strategies:
  1. Post-discharge care consultation
  2. Language Assessment
  3. Teach Back for Information and Skills
Other: Standard of Care (Reference) — No specific Transitional Care Strategy

SUMMARY:
Funded by the Patient Centered Outcome Research Institute (PCORI), nationally recognized leaders in health care and research methods are partnering with patients and caregivers to evaluate the effectiveness of current efforts at improving care transitions and develop recommendations on best practices for patient-centered care transitions and guidance for spreading them across the U.S.

DETAILED DESCRIPTION:
Patients in the U.S. suffer harm too often as they move between sites of health care, and their caregivers experience significant burden. Unfortunately, the usual approach to health care does not support continuity and coordination during such "care transitions" between hospitals, clinics, home or nursing homes. Poorly managed patient care transitions can lead to worsening symptoms, adverse effects from medications, unaddressed test results, failed follow-up testing, and excess rehospitalizations and ER visits.

Specific Aims:

1. Identify the transitional care outcomes and components that matter most to patients and caregivers.
2. Determine which evidence-based transitional care components (TCCs) or clusters most effectively yield patient and caregiver desired outcomes overall and among diverse patient and caregiver populations in different types of care settings and communities.
3. Identify barriers and facilitators to the implementation of specific TCCs or clusters of TCCs for different types of care settings and communities.
4. Develop recommendations for dissemination and implementation of the findings on the best evidence regarding how to achieve optimal TC services and outcomes for patients, caregivers and providers.

Study Design:

Capitalizing on the opportunity for a natural experiment observational study, the research team will conduct qualitative and quantitative studies. This 52-month study is divided into two distinct phases. During the first phase, Project ACHIEVE will use focus groups, with patients, caregivers, providers, and site visits to identify the transitional care outcomes and service components that matter most to patients. In this first phase, based on this information and an extensive evidence-based review of the research literature, the ACHIEVE team will develop surveys to be administrated in Phase II. The project team will conduct mail and phone surveys of patients and caregivers recruited from approximately 45 hospitals across the U.S. to assess what transitional care services patients and caregivers experience and how they are associated with outcomes. Additionally, the project team will conduct healthcare provider surveys and site visits to assess the facilitators and barriers to implementing transitional care strategies, organizational contexts (leadership and physician engagement, change culture, etc.), and community collaboration.

Outcomes and Impact:

Through rigorous study and evaluation, Project ACHIEVE will:

1. Identify best practices in care transitions that matter most to patients and their caregivers, and reduce excess emergency department and hospital utilization.
2. Develop a toolkit to guide informed decisions and spread these best practices across the U.S.
3. Develop Care Transitions Surveys that can standardize evaluation of patients' and caregivers' experience with care transitions.

ELIGIBILITY:
Inclusion Criteria:

* diverse high risk patient populations, including those with:

  1. multiple chronic conditions
  2. mental health issues
  3. rural area domicile
  4. limited English proficiency or low health literacy
  5. low socioeconomic status
  6. Medicare and Medicaid dual eligible
  7. disabled and younger than 65.

Exclusion Criteria:

* children
* non-Medicare patients
* Under police custody
* Under suicide watch
* In-hospital death
* Transferred (not discharged) to another acute care hospital
* Discharged against medical advice
* Admission for primary diagnosis of psychiatric conditions
* Admission for rehabilitation
* Admission for medical treatment of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Project ACHIEVE will focus on Medicare fee-for-services beneficiaries and study diverse high risk patient populations, including those with: 1) multiple chronic conditions; 2) mental health issues; 3) rural area domicile; 4) limited English proficiency or low health literacy; 5) low socioeconomic status; 6) Medicare and Medicaid dual eligible; 7) disabled and younger than 65.
Sampling Method: Probability Sample
Enrollment: 7939 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark V Williams, MD, Principal Investigator — University of Kentucky
Locations (1):
- UK Healthcare, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Brock J, Jack B, Mittman B, Naylor M, Sorra J, Mays G, Williams MV; Project ACHIEVE Team. Project ACHIEVE - using implementation research to guide the evaluation of transitional care effectiveness. BMC Health Serv Res. 2016 Feb 19;16:70. doi: 10.1186/s12913-016-1312-y. PMID 26896024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Any individual participant may have experienced more than one intervention.
Groups:
- Participants Receiving Transitional Care Strategies: Participants were exposed to one or more of five different transitional care strategies, or were part of a reference group that did not receive a specific transitional care strategy.
Period: Patient Communication and Care
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 2158
Completed | 2158
Not Completed | 0
Period: Home-Based Trust and Plain Language
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 1979
Completed | 1979
Not Completed | 0
Period: Hospital-Based Trust and Plain Language
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 2090
Completed | 2090
Not Completed | 0
Period: Patient/Family Caregiver Assessment
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 3093
Completed | 3093
Not Completed | 0
Period: Assessment and Teach Back
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 508
Completed | 508
Not Completed | 0
Period: Reference
Arm/Group | Participants Receiving Transitional Care Strategies
Started | 2042
Completed | 2042
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Recieving Transitional Care Strategies: Participants received one or more of 5 transitional care strategies, or were part of a reference group that received no specific transitional care strategy.
Arm/Group | Participants Recieving Transitional Care Strategies
Number analyzed (Participants) | 7939
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants may have experienced one or more interventions.
  Participants
    Patient Communication: number analyzed (Participants) | 2158
    Patient Communication: <=18 years | 0
    Patient Communication: Between 18 and 65 years | 337
    Patient Communication: >=65 years | 1821
    Home-Based Trust: number analyzed (Participants) | 1979
    Home-Based Trust: <=18 years | 0
    Home-Based Trust: Between 18 and 65 years | 200
    Home-Based Trust: >=65 years | 1779
    Hospital-Based Trust: number analyzed (Participants) | 2090
    Hospital-Based Trust: <=18 years | 0
    Hospital-Based Trust: Between 18 and 65 years | 172
    Hospital-Based Trust: >=65 years | 1918
    Patient/Family Caregiver Assessment: number analyzed (Participants) | 3093
    Patient/Family Caregiver Assessment: <=18 years | 0
    Patient/Family Caregiver Assessment: Between 18 and 65 years | 208
    Patient/Family Caregiver Assessment: >=65 years | 2885
    Assessement and Teach Back: number analyzed (Participants) | 508
    Assessement and Teach Back: <=18 years | 0
    Assessement and Teach Back: Between 18 and 65 years | 47
    Assessement and Teach Back: >=65 years | 461
    Reference: number analyzed (Participants) | 2042
    Reference: <=18 years | 0
    Reference: Between 18 and 65 years | 336
    Reference: >=65 years | 1706
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants may have received one or more transitional care strategies.
  years
    Patient Communication: number analyzed (Participants) | 2158
    Patient Communication | 70.50 (10.38)
    Home-Based Trust: number analyzed (Participants) | 1979
    Home-Based Trust | 72.04 (9.64)
    Hospital-Based Trust: number analyzed (Participants) | 2090
    Hospital-Based Trust | 72.62 (9.34)
    Patient/Family Caregiver Assessment: number analyzed (Participants) | 3093
    Patient/Family Caregiver Assessment | 73.55 (9.04)
    Assessment and Teach Back: number analyzed (Participants) | 508
    Assessment and Teach Back | 72.42 (8.91)
    Reference: number analyzed (Participants) | 2042
    Reference | 71.69 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants may have received one or more transitional care strategies.
  Participants
    Patient Communication: number analyzed (Participants) | 2158
    Patient Communication: Female | 1093
    Patient Communication: Male | 1065
    Home-Based Trust: number analyzed (Participants) | 1979
    Home-Based Trust: Female | 1102
    Home-Based Trust: Male | 877
    Hospital-Based Trust: number analyzed (Participants) | 2090
    Hospital-Based Trust: Female | 1082
    Hospital-Based Trust: Male | 1008
    Patient/Family Caregiver Assessment: number analyzed (Participants) | 3093
    Patient/Family Caregiver Assessment: Female | 1636
    Patient/Family Caregiver Assessment: Male | 1457
    Assessment and Teach Back: number analyzed (Participants) | 508
    Assessment and Teach Back: Female | 268
    Assessment and Teach Back: Male | 240
    Reference: number analyzed (Participants) | 2042
    Reference: Female | 1093
    Reference: Male | 949
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants may have received one or more transitional care strategies.
  Participants
    Patient Communication: number analyzed (Participants) | 2158
    Patient Communication: Hispanic or Latino | 243
    Patient Communication: Not Hispanic or Latino | 1809
    Patient Communication: Unknown or Not Reported | 106
    Home-Based Trust: number analyzed (Participants) | 1979
    Home-Based Trust: Hispanic or Latino | 250
    Home-Based Trust: Not Hispanic or Latino | 1627
    Home-Based Trust: Unknown or Not Reported | 102
    Hospital-Based Trust: number analyzed (Participants) | 2090
    Hospital-Based Trust: Hispanic or Latino | 445
    Hospital-Based Trust: Not Hispanic or Latino | 1539
    Hospital-Based Trust: Unknown or Not Reported | 106
    Patient/Family Caregive Assessment: number analyzed (Participants) | 3093
    Patient/Family Caregive Assessment: Hispanic or Latino | 580
    Patient/Family Caregive Assessment: Not Hispanic or Latino | 2345
    Patient/Family Caregive Assessment: Unknown or Not Reported | 168
    Assessment and Teach Back: number analyzed (Participants) | 508
    Assessment and Teach Back: Hispanic or Latino | 83
    Assessment and Teach Back: Not Hispanic or Latino | 394
    Assessment and Teach Back: Unknown or Not Reported | 31
    Reference: number analyzed (Participants) | 2042
    Reference: Hispanic or Latino | 229
    Reference: Not Hispanic or Latino | 1643
    Reference: Unknown or Not Reported | 170
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants may have received one or more transitional care strategies.
  Participants
    Patient Communication: number analyzed (Participants) | 2158
    Patient Communication: American Indian or Alaska Native | 21
    Patient Communication: Asian | 46
    Patient Communication: Native Hawaiian or Other Pacific Islander | 8
    Patient Communication: Black or African American | 141
    Patient Communication: White | 1702
    Patient Communication: More than one race | 41
    Patient Communication: Unknown or Not Reported | 199
    Home-Based Trust: number analyzed (Participants) | 1979
    Home-Based Trust: American Indian or Alaska Native | 12
    Home-Based Trust: Asian | 58
    Home-Based Trust: Native Hawaiian or Other Pacific Islander | 5
    Home-Based Trust: Black or African American | 234
    Home-Based Trust: White | 1449
    Home-Based Trust: More than one race | 38
    Home-Based Trust: Unknown or Not Reported | 183
    Hospital-Based Trust: number analyzed (Participants) | 2090
    Hospital-Based Trust: American Indian or Alaska Native | 21
    Hospital-Based Trust: Asian | 87
    Hospital-Based Trust: Native Hawaiian or Other Pacific Islander | 9
    Hospital-Based Trust: Black or African American | 155
    Hospital-Based Trust: White | 1504
    Hospital-Based Trust: More than one race | 28
    Hospital-Based Trust: Unknown or Not Reported | 286
    Patient/Family Caregiver Assessment: number analyzed (Participants) | 3093
    Patient/Family Caregiver Assessment: American Indian or Alaska Native | 28
    Patient/Family Caregiver Assessment: Asian | 122
    Patient/Family Caregiver Assessment: Native Hawaiian or Other Pacific Islander | 19
    Patient/Family Caregiver Assessment: Black or African American | 296
    Patient/Family Caregiver Assessment: White | 2144
    Patient/Family Caregiver Assessment: More than one race | 49
    Patient/Family Caregiver Assessment: Unknown or Not Reported | 435
    Assessment and Teachback: number analyzed (Participants) | 508
    Assessment and Teachback: American Indian or Alaska Native | 1
    Assessment and Teachback: Asian | 13
    Assessment and Teachback: Native Hawaiian or Other Pacific Islander | 1
    Assessment and Teachback: Black or African American | 60
    Assessment and Teachback: White | 362
    Assessment and Teachback: More than one race | 12
    Assessment and Teachback: Unknown or Not Reported | 59
    Reference: number analyzed (Participants) | 2042
    Reference: American Indian or Alaska Native | 15
    Reference: Asian | 37
    Reference: Native Hawaiian or Other Pacific Islander | 9
    Reference: Black or African American | 177
    Reference: White | 1577
    Reference: More than one race | 28
    Reference: Unknown or Not Reported | 199

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmission
Description: Readmission to the hospital within 30 days of discharge.
Time Frame: 30 days post hospital discharge
Population: Any individual participant may have experienced more than one group; therefore, the sum of participants across the arms exceeds the total sample size. Results data are shown for the entire arm (overall) and are also broken down into subgroups.
Measure: Number (95% Confidence Interval); unit: odds ratio
Groups:
- Patient Communication and Care Management: Participants received one more transitional care strategies.
  Patient Communication and Care Management: Received the following Transitional Care strategies:
  1. Helpful Health Care Contact OR Symptom Management
  2. Post-discharge Care Consultation
  3. Patient Goal/Preference Assessment
  4. Plain Language Communication in Hospital
  5. Plain Language Communication at Home
  6. Transition Summary for Patients and Family Caregivers
- Home-Based Trust, Plain Language, and Coordination: Participants received one more transitional care strategies.
  Home-Based Trust, Plain Language, and Coordination: Received the following Transitional Care Strategies:
  1. Transition Team
  2. Home visits
  3. Plain Language Communication at Home
  4. Promote Trust at Home
  5. Referral to Community Services
  6. Follow-up Appointment
- Hospital-Based Trust, Plain Language, and Coordination: Participants received one more transitional care strategies.
  Hospital-Based Trust, Plain Language, and Coordination: Received the following Transitional Care Strategies:
  1. Post-discharge care consultation
  2. Identify High-Risk Patients and Intervene
  3. Medication Reconciliation
  4. Plain Language Communication in Hospital
  5. Promote Trust in the Hospital
  6. Transition Summary for Patients and Family Caregivers
- Patient/Family Caregiver Assessment and Information Exchange a: Participants received one more transitional care strategies.
  Patient/Family Caregiver Assessment and Information Exchange among Providers: Received the following Transitional Care Strategies:
  1. Patient Goal/Preference Assessment
  2. Identify High-Risk Patients and Intervene
  3. Timely Exchange of Critical Patient Information among Providers
  4. Patient/Family Caregiver Transitional Care Needs Assessment
- Assessment and Teach Back: Participants received one more transitional care strategies.
  Assessment and Teach Back: Received the following Transitional Care Strategies:
  1. Post-discharge care consultation
  2. Language Assessment
  3. Teach Back for Information and Skills
- Reference: Participants were not involved in a specific transitional care strategy.
  Standard of Care: No specific Transitional Care Strategy
Arm/Group | Patient Communication and Care Management | Home-Based Trust, Plain Language, and Coordination | Hospital-Based Trust, Plain Language, and Coordination | Patient/Family Caregiver Assessment and Information Exchange a | Assessment and Teach Back | Reference
Number analyzed (Participants) | 2158 | 1979 | 2090 | 3093 | 508 | 2042
odds ratio
  Overall | .956 [.753 to 1.214] | .949 [.725 to 1.242] | .698 [.538 to .905] | .972 [.697 to 1.356] | 1.56 [.940 to 2.590] | .964 [.723 to 1.286]
  Multiple Chronic Conditions | .894 [.694 to 1.152] | .977 [.756 to 1.264] | .848 [.660 to 1.089] | 1.009 [.787 to 1.293] | 1.137 [.778 to 1.660] | .85 [.625 to 1.155]
  Mental Health Issues | 1.075 [.64 to 1.804] | .787 [.466 to 1.329] | .63 [.372 to 1.066] | .736 [.416 to 1.300] | 1.421 [.579 to 3.486] | .636 [.335 to 1.209]
  Rural Area Domicile | .885 [.479 to 1.635] | .776 [.455 to 1.325] | .777 [.435 to 1.387] | 1.021 [.511 to 2.039] | .122 [.013 to 1.159] | .665 [.334 to 1.325]
  Low Health Literacy | 1.113 [.776 to 1.595] | 1.129 [.771 to 1.652] | .681 [.471 to .984] | .916 [.603 to 1.392] | 1.057 [.575 to 1.941] | .927 [.610 to 1.409]
  Medicare/Medicaid Dual Eligible | 1.133 [.672 to 1.911] | .687 [.390 to 1.211] | .706 [.410 to 1.215] | .889 [.485 to 1.630] | 1.357 [.625 to 2.946] | .59 [.316 to 1.101]
  Disabled, <65 | 1.066 [.574 to 1.979] | .855 [.454 to 1.609] | .960 [.519 to 1.773] | 1.639 [.826 to 3.255] | 1.192 [.427 to 3.327] | 1.031 [.491 to 2.164]

2. Primary Outcome: Emergency Department (ED) Visit
Description: Visit to the ED within 30 days of hospital discharge.
Time Frame: 30 days post hospital discharge
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Patient Communication and Care Management | Home-Based Trust, Plain Language, and Coordination | Hospital-Based Trust, Plain Language, and Coordination | Patient/Family Caregiver Assessment and Information Exchange a | Assessment and Teach Back | Reference
Number analyzed (Participants) | 2158 | 1979 | 2090 | 3093 | 508 | 2042
Odds Ratio
  Overall | .946 [.787 to 1.137] | 1.031 [.839 to 1.266] | .803 [.657 to .981] | 1.091 [.834 to 1.428] | 1.524 [1.013 to 2.295] | .983 [.787 to 1.228]
  Multiple Chronic Conditions | .95 [.77 to 1.163] | 1.057 [.863 to 1.294] | .927 [.760 to 1.131] | 1.035 [.848 to 1.264] | .988 [.717 to 1.361] | .931 [.732 to 1.185]
  Mental Health Issues | 1.006 [.684 to 1.478] | .879 [.598 to 1.291] | .727 [.492 to 1.072] | 1.115 [.747 to 1.663] | 1.36 [.676 to 2.739] | .909 [.574 to 1.439]
  Rural Area Domicile | 1.013 [.601 to 1.708] | .756 [.491 to 1.163] | 1.392 [.755 to 2.566] | 1.082 [.578 to 2.026] | .246 [.032 to 1.874] | .798 [.445 to 1.429]
  Low Health Literacy | 1.125 [.855 to 1.480] | 1.097 [.829 to 1.452] | .867 [.656 to 1.147] | 1.099 [.819 to 1.473] | 1.086 [.673 to 1.753] | .939 [.682 to 1.293]
  Medicare/Medicaid Dual Eligible | .747 [.499 to 1.119] | .621 [.405 to .953] | .746 [.497 to 1.120] | .85 [.541 to 1.334] | .85 [.451 to 1.605] | .5 [.305 to .821]
  Disabled, <65 | .909 [.545 to 1.516] | .63 [.382 to 1.039] | .685 [.390 to 1.201] | .761 [.429 to 1.349] | 1.024 [.407 to 2.577] | .564 [.314 to 1.012]

ADVERSE EVENTS:
Time Frame: 30 days post hospital discharge
Description: Adverse events, serious adverse events, and all-cause mortality were not assessed as part of this study.
Arm/Group | Patient Communication and Care Management | Home-Based Trust, Plain Language, and Coordination | Hospital-Based Trust, Plain Language, and Coordination | Patient/Family Caregiver Assessment and Information Exchange a | Assessment and Teach Back | Reference
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02354482/Prot_SAP_000.pdf